CLINICAL TRIAL: NCT03124628
Title: Effects of Flywheel Resistance Exercise Training on Muscle and Walking Function in Teenagers and Young Adults With Cerebral Palsy
Brief Title: Effects of Flywheel Exercise on Muscle and Walking Function in Teenagers and Young Adults With Cerebral Palsy
Acronym: CP-Flywheel
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Rodrigo Fernandez Gonzalo, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Flywheel CP; 16037 (Other Grant/Funding Number: Promobilia)
Record Dates: First submitted 2017-03-17; First posted 2017-04-24 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flywheel resistance exercise (Experimental): During 8 weeks, all the subjects will follow a standard resistance exercise training program within the Stockholm Habilitation Center system. In addition, patients in this arm will perform flywheel leg press resistance exercise twice per week.
  Interventions: Other: Flywheel resistance exercise
- Weight-stack resistance exercise (Active Comparator): During 8 weeks, all the subjects will follow a standard resistance exercise training program within the Stockholm Habilitation Center system. In addition, patients in this arm will perform conventional, weight-stack leg press resistance exercise twice per week.
  Interventions: Other: Weight-stack resistance exercise

INTERVENTIONS:
Other: Flywheel resistance exercise — Flywheel resistance exercise, originally designed to maintain function, size and quality of skeletal muscle during spaceflight, employs iso-inertial technology rather than gravity dependent weights, which allows for coupled accommodated concentric and eccentric muscle actions, and brief episodes of eccentric overload.
  Other Names: Yo-Yo technology
  Arms: Flywheel resistance exercise
Other: Weight-stack resistance exercise — Conventional weight-stack resistance exercise
  Other Names: Conventional resistance exercise
  Arms: Weight-stack resistance exercise

SUMMARY:
The main purpose of this project is to improve physical function and muscle health in teenagers and young adults with cerebral palsy (CP) by using an eccentric-overload resistance exercise model

Specific aims

1. To compare the efficacy of eccentric-overload vs. weight stack resistance exercise in inducing muscle, functional and gait performance adaptations in teenagers with CP.
2. To increase force, power and muscle mass in the lower limbs of patients with cerebral palsy.
3. To improve gross motor function, balance and gait through eccentric-overload resistance exercise in teenagers suffering from cerebral palsy.

We hypothesize that the time-effective flywheel resistance exercise paradigm will result in greater gains in muscle mass and function in teenagers with CP, when compared with conventional weight-stack technology. Importantly, we believe these adaptations will be translated into enhanced gross motor function, balance and gait performance.

Forty teenagers and young adults (age range 16-23 yr) with spastic CP will be recruited. They will be randomly assigned to flywheel (FL; n=20) or weight-stack (WS; n=20) resistance exercise. During 8 weeks, all the teenagers will follow a standard resistance exercise training program within the Stockholm Habilitation Center system. In addition, patients will perform either flywheel (FL group) or conventional (WS group) leg press resistance exercise twice per week. Muscle force, power and activity (electromyography; EMG), leg extension lag, co-contraction, balance, functional mobility, gait quality, and muscle and fat thickness of lower extremities are assessed in all patients before and after the 8-week intervention (Fig. 1).

ELIGIBILITY:
Inclusion Criteria:

* Teenagers and young adults between 16-25 years of age
* Unilateral or bilateral spastic cerebral palsy
* Gross Motor Function Classification System (GMFCS) of level I, II or III.

Exclusion Criteria

* Surgical treatments of the knee extensor apparatus within the last 12 months
* Botulinum toxin treatment within the last six months
* Ongoing intrathecal baclofen treatment

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Muscle performance | Change from pre- to post-intervention (8 wks)
  Unilateral maximal voluntary isometric force is measured in both legs with force sensors. Similarly, unilateral (both legs) concentric and eccentric peak power is assessed through an encoder system. Furthermore, dynamic force during concentric and eccentric actions is measured via force sensors.
Muscle architecture | Change from pre- to post-intervention (8 wks)
  Vastus lateralis muscle thickness, together with fascicle pennation angle and muscle echogenicity, will be assessed using ultrasound technique in both legs. Thigh circumference will be assessed using measurement tape.
Electromyography of lower limb muscles | Change from pre- to post-intervention (8 wks)
  Muscle activation (mV) will be assessed in lower limb muscles (i.e. vastus lateralis, biceps femoris, gluteus medius, medial gastrocnemius) using surface electromyography techniques
Assessment of activities of daily living | Change from pre- to post-intervention (8 wks)
  Assessment of activities of daily living is measured using the Timed Up-and-Go test, the Chair-stand and the 6-min walking test.
Gait performance adaptations to training including muscle activation and co-contraction during walking | Change from pre- to post-intervention (8 wks)
  Gait performance will be analyzed using an 8-camera 3-D kinematic VICON system and force platforms at the Motion Analysis Laboratory, Astrid Lindgren Children's Hospital. Overall gait pathology will also be assessed using the multivariate Gait Deviation Index. Muscle activation and co-contraction during gait will be assessed using wireless surface electromyography
Gross motor function | Change from pre- to post-intervention (8 wks)
  Gross motor function will be assessed using Gross Motor Function Measure (GMFM)
Balance | Change from pre- to post-intervention (8 wks)
  Static and dynamic balance is assessed using force platforms at the Motion Analysis Laboratory, Astrid Lindgren Children's Hospital
Muscle spasticity | Change from pre- to post-intervention (8 wks)
  Spasticity will be assessed using the Ashworth scale

SECONDARY OUTCOMES:
Subcutaneous fat thickness | Change from pre- to post-intervention (8 wks)
  Subcutaneous fat thickness of the thigh of both legs will be assess using ultrasound techniques

CONTACTS AND LOCATIONS:
Overall Officials: Eva Pontén, MD, PhD, Study Director — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No